CLINICAL TRIAL: NCT04328311
Title: The Impact of Watermelon Juice on Blood Pressure in Young Healthy Adults
Brief Title: The Impact of Watermelon Juice on Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Charlotte E Mills, Lecturer, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 34/19
Record Dates: First submitted 2020-01-07; First posted 2020-03-31 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-01

CONDITIONS: Healthy Aging
Keywords: Watermelon; L-citrulline; Blood pressure
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Watermelon juice
  Interventions: Other: Watermelon Juice
- Control (Other): Low nitrate water.
  Interventions: Other: Water

INTERVENTIONS:
Other: Watermelon Juice — 500 mL watermelon juice (What a Melon), containing ~1 g of L-citrulline.
  Arms: Active
Other: Water — 500 mL low nitrate water
  Arms: Control

SUMMARY:
L-citrulline is found naturally in watermelon. Recently interest has increased for this amino acid due to potential health benefits. Notably, L-citrulline has the potential to lead to dilation of blood vessels due to its involvement in the production of nitric oxide.

The study will be an acute single blind, randomised controlled, crossover intervention study in healthy, young volunteers. Participants receive either the test watermelon drink or control drink (water). Blood samples and vascular measures (by a single-cuff based method) will be measured at baseline. Vascular measures will be repeated at 15-minute intervals between 0-2 hours and a second blood sample will be drawn at 1.5 hours to coincide with the estimated peak plasma L-citrulline. Citrulline, arginine and nitric oxide metabolites will be measured in the blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18-30 years
* Healthy (as per exclusion criteria)
* Able to understand information sheet
* Willing to comply with the study protocol
* Able to give informed consent.

Exclusion Criteria:

* Medical history of myocardial infarction
* Medical history of angina
* Medical history of thrombosis
* Medical history of stroke
* Medical history of cancer
* Medical history of high cholesterol
* Medical history of liver diseases
* Medical history of renal diseases
* Medical history of respiratory diseases
* Medical history of bowel diseases
* Medical history of diabetes
* Medical history of other endocrine disorders
* BMI <18.5 kg/m2 or >25 kg/m2
* Blood pressure <90/60 or > 140/90 mmHg
* Current use of antihypertensive medication
* Pregnant or lactating
* Alcohol intake > 14 units/week
* Cigarette smoker (or quit within the last 6 months)
* Vigorous exercise > 3 times/ week

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure | At baseline (t= 0 hours) and 15 minute intervals until t= 2 hours.
  Blood pressure by automated device

SECONDARY OUTCOMES:
Change in NOx (nitric oxide metabolites) | At baseline (t= 0 hours) and t=1.5 hours.
  Plasma nitrate and nitrite concentration
Change in l-arginine | At baseline (t= 0 hours) and t=1.5 hours.
  L-arginine concentration
Change in l-citrulline | At baseline (t= 0 hours) and t=1.5 hours.
  L-citrulline concentration

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No